CLINICAL TRIAL: NCT06240221
Title: A Clinical Registry to Track the Real World Use of the Saber-C® Cervical Fusion Device When Used for the Treatment of
Brief Title: A Clinical Registry to Track the Real World Use of the Saber-C® Cervical Fusion Device
Status: Enrolling by invitation | Type: Observational
Sponsor: Research Source (Network)
Responsible Party: Sponsor
Other Study IDs: Elevation Spine Reg-02
Record Dates: First submitted 2024-01-05; First posted 2024-02-02 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cervical Disc Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Saber-C: All enrolled patients will receive the Elevation Spine Saber-C System according to surgeon standard of care.
  Interventions: Device: Elevation Spine Saber-C System

INTERVENTIONS:
Device: Elevation Spine Saber-C System — Device: Elevation Spine Saber-C System Elevation Spine Saber-C System will be fixated between C2 through T1 according to surgeon standard of care at clinical practices through the United States.
  Other Names: Saber C, OVE, ODP, KWQ

SUMMARY:
The objective of this registry study is to collect radiographic and clinical outcome measures to determine the effectiveness of the Saber-C device.

DETAILED DESCRIPTION:
The purpose of this Clinical Registry is to track the real world use the Saber-C cervical fusion device when used for the treatment of Cervical Degenerative Disc Disease from C-2 to T1 for Anterior Cervical Discectomy and Fusion (ACDF). The registry is intended to profile the use of the Saber-C cervical fusion device when used according to surgeon standard of care at clinical practices throughout the United States. The focus of the registry will be to track and better understand the safety, effectiveness and market value of the Saber-C cervical fusion device.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Planned treatment with the Saber-C implant
* Subject is willing and able to sign informed consent

Exclusion Criteria:

* Subject is pregnant
* Subject is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A patient who meets all inclusion criteria and none exclusion criteria will be enrolled in the study. A patient is considered enrolled upon placement of the Elevation Spine Saber-C System during the surgical procedure. If the surgeon decides intra-operatively not to utilize Saber-C, the patient will be considered a screen failure.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Cervical spinal fusion status assessed via X-rays and CT scans | 1 year
  Cervical spinal fusion status will be assessed via X-rays and CT scans at 1 year post-surgery
Clinical outcome via neck visual analog scale (VAS) | 1 year
  Standard of care patient reported neck visual analog scale (VAS) will be used to evaluate patient pain. On a scale of 0 to 10 with a score of 0 being no pain and a score of 10 being worst pain. A low score means a better clinical outcome. A high score means a worse clinical outcome.
Clinical outcome via neck disability index (NDI) | 1 year
  Standard of care patient reported neck disability index (NDI) will be used to evaluate patient pain and quality of life. On a vertical scale of 0 to 5 with a score of 0 meaning neck pain (if any) does not interfere with life activities and 5 meaning neck pain strongly interferes with life activities. A low score means a better clinical outcome. A high score means a worse clinical outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Strenge Spine, Paducah, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No